CLINICAL TRIAL: NCT00420563
Title: A Phase II Randomized Study to Assess the Benefit of a Metronomic Chemotherapy by Cyclophosphamide Versus Megestrol in Palliative Cancer
Brief Title: Metronomic Chemotherapy by Cyclophosphamide Versus Megestrol in Palliative Cancer
Acronym: PALANGI-0601
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAL-ANGI 0601
Record Dates: First submitted 2007-01-09; First posted 2007-01-11 (Estimated); Last update posted 2012-07-23 (Estimated); Status verified 2012-07

CONDITIONS: Cancer
Keywords: Cancer, palliative treatment
MeSH Terms: conditions — Neoplasms | interventions — Cyclophosphamide; Megestrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CYCLOPHOSPHAMIDE (Experimental)
  Interventions: Drug: CYCLOPHOSPHAMIDE
- MEGESTROL (Active Comparator)
  Interventions: Drug: MEGESTROL

INTERVENTIONS:
Drug: CYCLOPHOSPHAMIDE — 50 mg x 2 /day , per os, nonstop until disease progression or toxicity or patient decision
  Arms: CYCLOPHOSPHAMIDE
Drug: MEGESTROL — 320 mg/day, per os, 2 pills of 160 mg one time, nonstop until disease progression or toxicity or patient decision
  Arms: MEGESTROL

SUMMARY:
The scope of the trial is to assess the free progression rate at 2 months for each group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18
* PS-WHO < or = 1
* Histologically proven cancer
* No other therapeutic proposal
* Treatment can be orally taken
* Radiologic proof of evolutive character of the disease
* Effective contraception

Exclusion Criteria:

* Hypercalcemia ( Ca > 2.65 mmol/l)
* Breast cancer
* Thrombosis or pulmonary embolism
* Dysphagia, malabsorption
* Polynuclear neutrophil leukocytes < 1000/mm3
* Treatment with Tegretol
* Active and uncontrolled infection
* Evolutive psychiatric disease
* Pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2006-09; Primary Completion 2009-01 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Progression free survival rate at 2 months | 2 months

SECONDARY OUTCOMES:
Progression free survival rate and objective response (RECIST) at 2, 4 and 6 months | After 2, 4 and 6 months of treatment
Toxicity according to NCI scale v3.0 | During study treatment
Biological markers | the 2 first months of treatment
Overall survival | Until death of the patient or until study analysis
Median time between the beginning of treatment and hospitalization due to progression or toxicity | time of the study

CONTACTS AND LOCATIONS:
Overall Officials: PENEL Nicolas, MD, Principal Investigator — Centre Oscar Lambret
Locations (4):
- France (4):
  - Centre Oscar Lambret, Lille
  - Hopital Saint Vincent, Lille
  - Centre Hospitalier Regional - Dermatology, Lille
  - Centre Hospitalier Regional - Oncology, Lille